CLINICAL TRIAL: NCT07373808
Title: Efficacy of Sciatic Nerve Electrical Stimulation and Therapeutic Exercise in the Management of Low-back Related Leg Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Ilustre Colegio Profesional de Fisioterapeutas de la Comunidad de Madrid (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25/504-E
Record Dates: First submitted 2025-11-25; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11

CONDITIONS: Sciatica
MeSH Terms: conditions — Sciatica | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Real PENS + Placebo TENS (Experimental): Participants will receive real ultrasound-guided dry needle insertion (0.30 mm × 60 mm and 0.30 mm ×50 mm) to the perineural region adjacent to the sciatic nerve at both the subgluteal fold and the posterior thigh (junction between the middle and distal thirds). Electrical stimulation will be applied using the Endomed 484® electrotherapy unit (PRIM Physio, Madrid, Spain) in continuous biphasic mode at low frequency (2 Hz), 250 μs pulse width for 30 minutes. Intensity will be adjusted to elicit a visible, mild muscle contraction.
  Simultaneously, adhesive electrodes will be placed near the intervention site but connected to a disabled channel to simulate placebo TENS.
  Interventions: Procedure: Percutaneous Electrical Nerve Stimulation; Procedure: Placebo Transcutaneous Electrical Nerve Stimulation; Procedure: Progressive Therapeutic Exercise Program
- Real TENS + Placebo PENS (Active Comparator): Participants will receive real superficial electrical stimulation via adhesive electrodes connected to the Endomed 484® unit, configured for TENS (non-invasive). Parameters will match those from Group 1 (continuous biphasic current, 2 Hz, 250 μs, 30 min), producing a clear sensory perception and mild muscle contraction.
  Simultaneously, a sham ultrasound-guided dry needling procedure will be performed using Streitberger placebo needles, which contact the skin superficially without penetration. Cables for PENS will be placed on the skin but connected to a disabled channel to simulate placebo PENS.
  Interventions: Procedure: Transcutaneous Electrical Nerve Stimulation; Procedure: Placebo Percutaneous Electrical Nerve Stimulation; Procedure: Progressive Therapeutic Exercise Program
- Real Dry Needling (without PENS) + Placebo TENS (Active Comparator): Participants will receive real ultrasound-guided dry needling as in Group 1 but without electrical stimulation. The needles will remain in place for 30 minutes, with the PENS channel disabled to act as placebo.
  Simultaneously, adhesive electrodes will be placed as in Group 1, with TENS channels disabled. Participants will be told the current is below the sensory threshold.
  The design of this intervention group aims to determine whether the therapeutic effects observed with the PENS technique are exclusively due to needle insertion (dry needling) or whether the passage of electrical current through the needle (as in Group 1) plays a decisive role in the outcomes obtained. To this end, real ultrasound-guided dry needling is applied at the same anatomical locations, but without activation of the electrical stimulation channel, the latter acting as a placebo. This comparison will allow the specific effect of electrical stimulation to be isolated within the context of the intervention.
  Interventions: Procedure: Placebo Transcutaneous Electrical Nerve Stimulation; Procedure: Real Dry Needling (without Percutaneous Electrical Nerve Stimulation); Procedure: Progressive Therapeutic Exercise Program
- Placebo PENS + Placebo TENS (Placebo Comparator): Participants will receive only sham interventions. Placebo PENS will be simulated with Streitberger needles (skin contact without penetration) and cable placement, and placebo TENS with adhesive electrodes connected to a disabled channel. Participants will be informed that current is below the sensory threshold. The procedure will last 30 minutes.
  Interventions: Procedure: Placebo Transcutaneous Electrical Nerve Stimulation; Procedure: Placebo Percutaneous Electrical Nerve Stimulation; Procedure: Progressive Therapeutic Exercise Program

INTERVENTIONS:
Procedure: Percutaneous Electrical Nerve Stimulation — Participants will receive real ultrasound-guided dry needle insertion (0.30 mm × 60 mm and 0.30 mm ×50 mm) to the perineural region adjacent to the sciatic nerve at both the subgluteal fold and the posterior thigh (junction between the middle and distal thirds). Electrical stimulation will be applied using the Endomed 484® electrotherapy unit (PRIM Physio, Madrid, Spain) in continuous biphasic mode at low frequency (2 Hz), 250 μs pulse width for 30 minutes. Intensity will be adjusted to elicit a visible, mild muscle contraction.
  Other Names: PENS
  Arms: Real PENS + Placebo TENS
Procedure: Placebo Transcutaneous Electrical Nerve Stimulation — Adhesive electrodes will be placed near the intervention site (sciatic nerve between the subgluteal fold and the distal third of the thigh) but connected to a disabled channel to simulate placebo TENS.
  Other Names: Placebo TENS
  Arms: Placebo PENS + Placebo TENS; Real Dry Needling (without PENS) + Placebo TENS; Real PENS + Placebo TENS
Procedure: Transcutaneous Electrical Nerve Stimulation — Participants will receive real superficial electrical stimulation via adhesive electrodes connected to the Endomed 484® unit, configured for TENS (non-invasive). Parameters will include continuous biphasic current, 2 Hz, 250 μs, 30 min, producing a clear sensory perception and mild muscle contraction.
  Other Names: TENS
  Arms: Real TENS + Placebo PENS
Procedure: Placebo Percutaneous Electrical Nerve Stimulation — A sham ultrasound-guided dry needling procedure will be performed using Streitberger placebo needles, which contact the skin superficially without penetration. Cables for PENS will be placed on the skin but connected to a disabled channel to simulate placebo PENS.
  Other Names: Placebo PENS
  Arms: Placebo PENS + Placebo TENS; Real TENS + Placebo PENS
Procedure: Real Dry Needling (without Percutaneous Electrical Nerve Stimulation) — Participants will receive real ultrasound-guided dry needling but without electrical stimulation. The needles will remain in place for 30 minutes, with the PENS channel disabled to act as placebo.
  Other Names: Real Dry Needling (without PENS)
  Arms: Real Dry Needling (without PENS) + Placebo TENS
Procedure: Progressive Therapeutic Exercise Program — The program will include five lumbopelvic strengthening and stabilization exercises plus a squat exercise. Each participant will attend one supervised weekly session led by a physiotherapist and will be encouraged to repeat the program at home at least twice a week. Progression will depend on pain tolerance and perceived exertion. Each session will include warm-up (5-7 min), strengthening (20-25min) and cool-down (5 min).
  Before starting with the main exercises, participants will do a warm-up designed to improve general and specific mobility of the lumbar spine and lower limbs, including five exercises (1 minute each). Then, strengthening exercises will be performed, including Curl-up, Bird-Dog, Side plank, Front plank, Glute bridge and Controlled partial squat. Finally, a brief cool-down period will be carried out, focused on active mobility and gentle stretching to facilitate recovery and reduce potential muscle overload, consisting of four exercises (1 minute each).

SUMMARY:
This clinical study focuses on people who experience long-term low-back related leg pain (commonly called sciatica). This type of pain is often associated with nerve irritation or compression in the lower spine and can cause symptoms like shooting or burning pain, tingling, numbness, or weakness in the leg. Many patients continue to suffer from this problem for months or years, and available treatments (including painkillers, anti-inflammatory drugs, or even surgery) do not always provide lasting relief. Because of this, there is a strong need to explore safe, non-drug, non-surgical therapies. The purpose of this study is to test the efficacy and safety of a treatment called Percutaneous Electrical Nerve Stimulation (PENS) when applied near the sciatic nerve, the large nerve that runs from the lower back through the buttock and down the leg, in combination with a therapeutic exercise program. PENS uses very thin sterile needles inserted under ultrasound guidance next to the nerve. A gentle electrical current is then applied for about 30 minutes to stimulate the nerve in a controlled way. This may help calm down nerve sensitivity, reduce inflammation, and decrease pain. We will compare PENS with three other options: Transcutaneous Electrical Nerve Stimulation (TENS): A commonly used therapy where mild electrical stimulation is applied through adhesive patches placed on the skin; Dry needling without electrical current: Thin needles are inserted under ultrasound guidance but no current is applied; and placebo treatment: A simulated version of the therapy with no active current, designed to look and feel similar so that participants do not know which treatment they are receiving. In addition to these treatments, all participants will take part in a structured exercise program aimed at strengthening the lower back, pelvis, and legs. Exercises like curl-ups, planks, bridges, bird-dogs, and squats will be supervised weekly for six weeks, with guidance to continue practicing at home. Exercise is included because it is known to help improve mobility, strength, and recovery in people with back problems. The study is designed as a randomized, controlled, double-blind trial, which means that participants are assigned to one of the four groups by chance (like flipping a coin), and neither the patients nor the therapists who collect the measurements will know which treatment has been given. This design ensures fairness and reliability of the results. We will measure: Back and leg pain levels, using a simple 0-10 scale; Disability, meaning how much the pain limits daily activities, measured with a well-known questionnaire; Quality of life, both physical and mental health aspects; Nerve-related pain features, like burning or electric-like sensations; and patients' global impression of improvement and any side effects. Assessments will take place before starting the treatment, at the end of the 6-week program, and then again at 3 and 6 months. This allows us to see both the short-, mid- and long-term effects. Safety considerations: Previous research shows that PENS and similar techniques are generally very safe. The most common side effects are mild and short-lasting, including temporary soreness, heaviness in the leg, or a small bruise. Serious complications are extremely rare. To minimize risks, all procedures will be carried out by experienced physiotherapists, using real-time ultrasound to guide needle placement and ensure accuracy. Only sterile, single-use needles are employed. By comparing PENS, TENS, dry needling, and placebo, this study seeks to determine whether PENS in combination with therapeutic exercise provides superior benefits in reducing pain, improving function, and enhancing quality of life for patients with sciatica-type low back pain. If successful, this treatment could become a valuable alternative to drugs or surgery, offering patients a safe and effective therapy to better manage their condition and regain daily function.

ELIGIBILITY:
Inclusion Criteria:

* Neuropathic-like LBRLP (sciatica).
* S-LANSS score ≥ 12 points.
* LBRLP lasting more than 6 months.
* Age between 18 and 70 years.
* LBRLP in the past 4 weeks has been severe enough to limit usual activities or change daily routines for more than 1 day.
* At least one period of 6 months to 1 year during which the participant did not go a full month without LBRLP.
* LBRLP intensity of at least 3/10 on the NPRS.
* Ability to provide informed consent.

Exclusion Criteria:

* Acute injury or recent major trauma history.
* Relevant painful conditions of the hip joint or pelvic/sacroiliac region.
* Symptoms compatible with cauda equina syndrome (loss of bladder/bowel control, sexual dysfunction, paralysis of lower limbs, etc.).
* Previous surgery on the spine, pelvis or hip.
* Prior treatment with anesthetic or anti-inflammatory blocks or with radiofrequency (facet, sacroiliac, radicular, epidural, etc.) in the past two years.
* Any neurological or systemic disease that could limit participation in the study.
* Inability to communicate in Spanish or understand study instructions and content.
* General contraindications for invasive physiotherapy and electrotherapy techniques.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline, 1 week post-intervention, and 3 and 6 months after the intervention.
  Pain intensity will be assessed using the NPRS, a single 11-point numerical rating scale widely validated across different patient populations, where 0 represents no pain and 10 represents the worst possible pain. Data obtained through the NPRS are easy to document, intuitively interpretable and meet regulatory requirements for pain assessment and documentation. The NPRS has been shown to be reliable in assessing LBP intensity, also predicting the degree of disability in these patients. A change of 2 points on the NPRS has been considered to reflect the MCID in patients with LBP, indicating that any change equal to or greater than this value can be considered clinically relevant. However, the MCID has not yet been established in patients with LBRLP and neuropathic characteristics; therefore, a variation of 2 points will be used as a reference value, as in patients with LBP and those with chronic pain in general.

SECONDARY OUTCOMES:
Disability | Baseline, 1 week post-intervention, and 3 and 6 months after the intervention.
  Disability will be assessed using the Oswestry Disability Index (ODI), an instrument designed to evaluate the degree of disability associated with acute, subacute and chronic LBP. The ODI consists of a total of 10 items, one assessing pain and the remaining nine assessing activities of daily living, each rated on a 6-point ordinal scale ranging from the best to the worst scenario (0-5 points). The scores for each item will be summed to obtain a total between 0 and 50 points, with the following categories: no disability (0-4 points), mild disability (5-14 points), moderate disability (15-24 points), severe disability (25-34 points) and complete disability (35-50 points). The ODI has been shown to be reliable and valid for assessing disability in patients with LBP and has been validated in Spanish. The MCID varies across studies; in this case, the smallest reported value (a change of 5 points) will be used as the reference for significant changes.
Health-related quality of life | Baseline, 1 week post-intervention, and 3 and 6 months after the intervention.
  The SF-12 questionnaire, a shortened version of the SF-36, will be used for this assessment. The SF-12 consists of 12 items that evaluate eight different parameters: physical functioning, role limitations due to physical problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems and mental health perception. The items are combined and transformed to provide both a physical and a mental health score, each ranging from 0 (worst) to 100 (best). The SF-12 has been shown to be valid and reliable in populations with chronic LBP. The MCID related to quality of life in patients with LBP has been established as improvements greater than 3.77 points in the mental component and 3.29 points in the physical component.
Neuropathic component of pain | Baseline, 1 week post-intervention, and 3 and 6 months after the intervention.
  This variable will be measured using the S-LANSS pain scale, a self-administered instrument designed to identify patients with pain of neuropathic characteristics. It is a simple scale consisting of seven items with binary responses (yes or no), relating to the presence of symptoms (five items) or clinical signs (two items). The maximum possible score is 24 points, with scores equal to or greater than 12 considered clear indicators of the presence of a neuropathic pain component. The S-LANSS scale has been shown to be reliable for diagnosing pain with neuropathic characteristics and has been validated in Spanish.
Global perceived improvement | 1 week post-intervention, and 3 and 6 months after the intervention.
  Global perceived improvement will be measured using a 7-point Likert scale ranging from "much worse" to "much better." Clinical improvement will be considered in participants who report feeling "moderately better" or "much better".
Adverse events | Through study completion, an average of 2 years.
  Adverse events will be defined as any problem related to the intervention that causes symptoms lasting at least two days or requiring specific treatment.

OTHER OUTCOMES:
Sociodemographic variables | Baseline.
  Sociodemographic data will be collected using a standardized form in which participants will be required to provide their age, gender, occupation, height, weight, ethnicity, education level, comorbidities, history of sports activity, symptoms in other joints, duration of symptoms and medication use.